CLINICAL TRIAL: NCT00589680
Title: Compliance With American Diabetes Association Treatment Guidelines for Adult Ketoacidosis
Status: Completed | Type: Observational
Sponsor: Marshall University (Other)
Responsible Party: Principal Investigator, Sharon Jones, Clinical Coordinator, Marshall University
Other Study IDs: 9137
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Diabetic Ketoacidosis
Keywords: Acidosis, Diabetic; Diabetic Acidosis; Diabetic Ketosis; Ketoacidosis, Diabetic; Ketosis, Diabetic
MeSH Terms: conditions — Diabetic Ketoacidosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 2: Patients treated for DKA under DKA protocol implemented by hospital
- 1: To establish a baseline on how patients are being treating with DKA in general and without a standardized DKA protocol

SUMMARY:
At this time, Saint Mary's Medical Center is currently in the process of implementing a standardized diabetic ketoacidosis (DKA) protocol. The first main goal of this project will be to evaluate patient outcomes to determine the effects of treating patients without a standardized protocol and to establish a baseline on how patients are being treating with DKA. The final goal of the project will be to compare outcomes of those patients not placed on the protocol to those that were treated using SMMC newly implemented DKA protocol. The overall goal of this project is to determine the benefit of an institutional DKA protocol.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to St. Mary's Medical Center with DKA
* >/= 18 years of age

Exclusion Criteria:

* < 18 years of age

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those patients admitted to St. Mary's Medical Center with a diagnosis of DKA.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay | Time in hospital

SECONDARY OUTCOMES:
ICU length of stay | hospital stay
ICU length of stay Hypoglycemic events (BG<60) | hospital stay
Time to correction of glucose level and anion gap | hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Jones, Pharm.D., Principal Investigator — St. Mary's Medical Center
Locations (1):
- St. Mary's Medical Center, Huntington, West Virginia, United States